CLINICAL TRIAL: NCT07183618
Title: Impact of Mental Training on the Stress of Anaesthesiology Residents Before Performing Obstetrical Epidural Analgesia: a Prospective Randomized Educational Trial
Brief Title: Impact of Mental Training on the Stress of Anaesthesiology Residents Before Performing Obstetrical Epidural Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Principal Investigator, jean.selim, Professor, University Hospital, Rouen
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: E2024-05
Record Dates: First submitted 2025-09-12; First posted 2025-09-19 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Medical Education; Resident Education; Anesthesia; Epidural Analgesia, Obstetric
Keywords: anesthesia residency; mental training; obstetrical epidural anesthesia; medical education

STUDY DESIGN:
Intervention Model Description: Residents were randomly assigned to either a "Control" group or a "Mental Training" group, the latter undergoing a mental preparation session before performing lumbar epidural anaesthesia. Randomisation was performed in blocks of eight by an external party and stratified by training year (second or third) and gender. Residents were informed they would be participating in a training session involving anaesthetic practice on a low-fidelity simulator.
  On the day of the simulation, residents were individually welcomed in a briefing room by an anaesthetist specialised in mental preparation. Group assignment was revealed from a sealed envelope and residents were informed that the simulation would involve acting as the on-call anaesthesia resident in a maternity ward. The scenario began with a call from a midwife requesting an epidural placement for a laboring patient. Depending on their assigned group, residents either received a mental preparation session or proceeded without it.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (no mental training) (No Intervention): Residents in the control group did not undergo any mental training prior to performing epidural placement.
- Mental training group (Experimental): Mental Training Group: Residents in the "Mental Training" group received a mental preparation session led by an anaesthesia physician qualified in medical pedagogy. Inspired by the "Breathe, Talk, See, Focus" procedure
  Interventions: Procedure: Mental training group

INTERVENTIONS:
Procedure: Mental training group — Mental Training Group: Residents in the "Mental Training" group received a mental preparation session led by an anaesthesia physician qualified in medical pedagogy. Inspired by the "Breathe, Talk, See, Focus" procedure
  Arms: Mental training group

SUMMARY:
Anaesthetists are trained from the beginning of their residency to perform high-risk procedures, often in high-stress environments, that can adversely affect both their technical and non-technical performance. Effective stress management is therefore essential, particularly before executing technical procedures. Recently, mental training has been introduced in the education of surgical residents to enhance performance under pressure. This study aimed to assess, using simulation, the impact of mental preparation on stress levels among anaesthesia residents before performing obstetric epidural analgesia.

DETAILED DESCRIPTION:
Residents were randomly assigned to either a "Control" group or a "Mental Training" group, the latter undergoing a mental preparation session before performing lumbar epidural anaesthesia. Randomisation was performed in blocks of eight by an external party and stratified by training year (second or third) and gender. Residents were informed they would be participating in a training session involving anaesthetic practice on a low-fidelity simulator.

On the day of the simulation, residents were individually welcomed in a briefing room by an anaesthetist specialised in mental preparation. Group assignment was revealed from a sealed envelope and residents were informed that the simulation would involve acting as the on-call anaesthesia resident in a maternity ward. The scenario began with a call from a midwife requesting an epidural placement for a laboring patient. Depending on their assigned group, residents either received a mental preparation session or proceeded without it. Both groups participated in a ten-minute briefing session.

ELIGIBILITY:
Inclusion Criteria: Eligible subjects for this study were anaesthesia and intensive care residents enrolled at the Faculty of Medicine and Pharmacy in Rouen. Residents were eligible if they were in the early stages of training (second and third years of residency) and had previously performed lumbar epidural anaesthesia multiple times in a maternity setting.

Exclusion Criteria: Exclusion criteria included first-year residents, as not all had performed obstetric lumbar epidural anaesthesia at the time of the study, and senior residents (fourth and fifth years).

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-02-28 (Actual)

PRIMARY OUTCOMES:
Comparison of the stress levels before and after performing obstetric epidural anaesthesia between residents who received mental preparation and those who did not. | Immediately after the simulation
  Thestress level was evaluated using the State-Trait Anxiety Inventory 6 (STAI-6) score

SECONDARY OUTCOMES:
Technical performance evaluation | During the simulation
  Technical performance was assessed with a validated checklist
Non-technical skills evaluation | During the simulation
  Non-technical skills was measured by the Anaesthetists' Non-Technical Skills (ANTS) score
Mental imagery abilities evaluation | Immediatly after the simulation
  Mental imagery abilities was assessed via the Mental Imagery Questionnaire
Residents' satisfaction score | Immediatly after the simulation
  Satisfaction score ranging from 0 to 10

CONTACTS AND LOCATIONS:
Locations (1):
- Rouen University Hospital, Rouen, Normandy, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fluteau L, Bourdon-Castel S, Kallout J, Lefevre-Scelles A, Sibert L, Besnier E, Clavier T, Compere V, Selim J. Impact of Mental Training on the stress of anaesthesiology residents before performing obstetrical epidural analgesia: a prospective randomised educational trial. Anaesth Crit Care Pain Med. 2025 Nov 15:101675. doi: 10.1016/j.accpm.2025.101675. Online ahead of print. PMID 41248877